CLINICAL TRIAL: NCT04306042
Title: A Survival Observational Study in Patients With Advanced IIIB-IV Squamous Cell Lung Cancer Receiving PD-1 Combination With Chemotherapy (RESPONSE)
Brief Title: A Survival Observational Study in Patients With Advanced IIIB-IV Squamous Cell Lung Cancer Receiving PD-1 Combination With Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Other Study IDs: CTONG1904
Record Dates: First submitted 2020-02-11; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Lung Squamous Cell Carcinoma Stage IV
MeSH Terms: interventions — Nivolumab; pembrolizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment: Patients diagnosed with primary stage IIIB-IV squamous cell lung cancer and treated in 92 medical centers between 01 September 2019 and 30 June 2020 will be targeted for study inclusion.
  Interventions: Drug: Nivolumab or Pembrolizumab

INTERVENTIONS:
Drug: Nivolumab or Pembrolizumab — Nivolumab or Pembrolizumab

SUMMARY:
This is a multi-center, open-label, non-interventional, retrospective registry study, with no pre-set statistical assumptions and will not intervene subject's clinical treatment or clinical management.

In the study, the clinical data of the subjects will be retrospectively collected from the electronic health records (EHR) of each research center. The clinical information will be based on the actual medical records of the cases. After the retrospective study time (June 30, 2020), patients will be followed for one-year and two-year survival. Clinical treatment and management will be based on local clinical practices and regulations. This study will record the actual diagnosis and treatment, and will not interfere with any clinical decision.

After subject-out, patients will be followed for one-year and two-year survivals, thus the follow-up consent will be exempted. All patients receiving PD-1 monoclonal antibody in combination with chemotherapy will be visited during the entire study period. At the end of study, investigator will check up on the conditions of patients who withdraw from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Men and woman, aged over 18
2. Cytology or histologically confirmed squamous cell lung cancer
3. Advanced squamous cell lung cancer, Stage IIIb to IV according to AJCC staging (version 8)
4. Patients receiving approved PD-1 mAb in combination with chemotherapy according to their condition
5. Patients receiving PD-1 mAb in combination with chemotherapy for at least one cycle (21 days)
6. Have imaging results with measurable tumor 2 weeks before receiving PD-1 mAb in combination with chemotherapy
7. Able to understand and comply with the requirements of the consent and voluntarily participate in the study

Exclusion Criteria:

1. Patients participating in other clinical studies
2. Severe medical data missing
3. Unable to understand the purpose of the study or not agree with the requirement of the study
4. Malignancies other than squamous cell lung cancer, history of malignancies
5. Unsuitable for the study according to investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with primary stage IIIB-IV squamous cell lung cancer and treated in 92 medical centers.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
2 year survival rate | 2 years
objective response rate | 2 years
disease control rate | 2 years
  free survival
median progression free survival | 2 years

SECONDARY OUTCOMES:
incidence of adverse reactions | 2 years
  Safety of the combination of PD-1 and chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Patients information without identification data will be shared within centers enrolled in the study to perform the data analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code